CLINICAL TRIAL: NCT06049940
Title: Randomized, Double-blind, Controlled Phase Ⅰ and Phase Ⅲ Clinical Trial to Evaluate the Safety and Immunogenicity of Tetanus Vaccine, Adsorbed in 18~44 Years Old Population
Brief Title: Safety and Immunogenicity of Tetanus Vaccine, Adsorbed in 18~44 Years Old Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-TT-3001
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Tetanus
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 630 Participants (including 30 subjects in phaseⅠ, 600 subjects in phase Ⅲ ) will receive one dose of experimental vaccine or control vaccine.
  Interventions: Biological: Investigational tetanus vaccine, adsorbed
- Control Group (Active Comparator): 630 Participants (including 30 subjects in phaseⅠ, 600 subjects in phase Ⅲ ) will receive one dose of experimental vaccine or control vaccine.
  Interventions: Biological: Control tetanus vaccine, adsorbed

INTERVENTIONS:
Biological: Investigational tetanus vaccine, adsorbed — The investigational vaccine was manufactured by Sinovac Life Sciences Co., Ltd. There is not less than 40IU tetanus toxoid in 0.5ml per dose.
  Arms: Experimental Group
Biological: Control tetanus vaccine, adsorbed — The control tetanus vaccine, adsorbed was manufactured by Chengdu Olymvax Biopharmaceuticals Inc.There is not less than 40IU tetanus toxoid in 0.5ml per dose.
  Arms: Control Group

SUMMARY:
This is a randomized, double-blind, positive controlled design clinical trial of tetanus vaccine, adsorbed manufactured by Sinovac Life Sciences Co., Ltd.The purpose of this study is to evaluate the safety and immunogenicity of tetanus vaccine, adsorbed in 18~44 years old population.

DETAILED DESCRIPTION:
This is a randomized, double-blind, positive controlled design clinical trial of tetanus vaccine, adsorbed.The purpose of this study is to evaluate the safety and immunogenicity of tetanus vaccine, adsorbed in 18~44 years old population.The study will conduct in two phases.A total of 1260 subjects including 60 subjects in phase Ⅰ and 1200 subjects in phase III will be enrolled.All of subjects in phase Ⅰ and phase III will be randomly assigned 2 groups in a 1:1 ratio to receive one dose of experimental vaccine or control vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy aldults aged 18-44 months;
* Proven legal identity;
* Subjects have the ability to understand and agree to sign the informed consent form.

Exclusion Criteria:

* Armpit temperature of persons with fever on the day of experimental vaccine administration>37.0 ℃;
* Previous history of tetanus infection;
* Has received tetanus vaccines or vaccines containing tetanus toxoid antigen (DTP, DTP, meningococcal conjugate vaccine, etc.) within the last 10 years, or has received a tetanus immunoglobulin or tetanus antitoxin within the previous 6 months;
* Women who are lactating, pregnant (with a positive urine pregnancy test) or planning to become pregnant within the last 3 months;
* History of asthma, allergy to vaccines or vaccine components, and severe adverse reactions to vaccines, such as urticaria, dyspnea, angioedema, or abdominal pain;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Have congenital or acquired immunodeficiency such as HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), juvenile rheumatoid arthritis (JRA);
* Thyroid disease or history of thyroidectomy, asplenia, functional asplenia, asplenia or splenectomy resulting from any condition;
* Severe chronic diseases,such as severe cardiovascular diseases, hypertension(Systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg) and diabetes that cannot be controlled by drugs, liver or kidney diseases,malignant tumors, etc;
* Currently suffering from or have suffered from encephalopathy (such as congenital brain hypoplasia, brain trauma, brain tumor, cerebral hemorrhage, cerebral infarction, brain infection, chemical poisoning, etc.); A history of convulsions, epilepsy, psychosis or a family history of psychosis, and other serious neurological disorders;
* Diagnosed abnormal blood coagulation function (e.g. coagulation factor deficiency, coagulation disorders, abnormal platelets) or obvious bruising or coagulation disorders;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* A long history of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Acute onset of various acute diseases or chronic diseases in the last 7 days;
* Participating in clinical studies of other vaccines or drugs;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1260 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions | within 30 days after vaccination
  Incidence of adverse reactions within 30 days after vaccination.
Incidence of local or systemic adverse reactions | Within 7 days after vaccination
  Incidence of local or systemic adverse reactions within 7 days after vaccination.
Incidence of grade 3 and above adverse reactions | Within 30 days after vaccination
  Incidence of grade 3 and above adverse reactions within 30 days after vaccination
Incidence of SAE related to vaccination | From the beginning of vaccination to 6 months after vaccination
  Incidence of SAE related to vaccination from the beginning of vaccination to 6 months after vaccination.

SECONDARY OUTCOMES:
The seroprotective rate of anti-tetanus toxiod antibody | 30 days after vaccination
  The seroprotective rate of anti-tetanus toxiod antibody 30 days after vaccination.
Long-term seroprotective rate of anti-tetanus toxiod antibody | 30 days after vaccination
  Long-term seroprotective rate of anti-tetanus toxiod antibody 30 days after vaccination.
Seroconversion rate of anti-tetanus toxiod antibody | 30 days after vaccination
  Seroconversion rate of anti-tetanus toxiod antibody 30 days after vaccination.
GMC of anti-tetanus toxiod antibody | 30 days after vaccination
  GMC of anti-tetanus toxiod antibody 30 days after vaccination.
GMC increase folds (GMI) of anti-tetanus toxiod antibody | 30 days after vaccination
  GMC increase folds (GMI) of anti-tetanus toxiod antibody 30 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqing Xie, Principal Investigator — Henan Provincial Center for Disease Prevention and Control
Locations (1):
- Liangyuan District Center for Disease Control and Prevention, Shangqiu, Henan, China